CLINICAL TRIAL: NCT06376279
Title: Genetisk Diagnostik Vid medfödda Metabola Sjukdomar
Brief Title: Genetic Diagnosis in Inborn Errors of Metabolism
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/351-31
Record Dates: First submitted 2024-01-29; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-01

CONDITIONS: Metabolic Disease; Mitochondrial Diseases; Epilepsy in Children; Epilepsy; LHON; Motor Neuron Disease
MeSH Terms: conditions — Metabolic Diseases; Mitochondrial Diseases; Epilepsy; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Muscle biopsy, skin biopsy, fibroblasts, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: IEM-EP — Data from IEM-inborn error of metabolism cohort of individuals

SUMMARY:
Inborn Errors of metabolism comprise a large number of rare conditions with a collective incidence of around 1/2000 newborns. Many disorders are treatable provided that a correct diagnosis can be established in time, and for many diseases novel therapies are being developed. Without treatment, many of the conditions result in early death or severe irreversible handicaps.

The Centre for Inherited Metabolic Diseases, CMMS at Karolinska university hospital, is an integrated expert center where clinical specialists work closely together with experts in laboratory medicine, combining clinical genetics, clinical chemistry, pediatrics, neurology, and endocrinology. The center serves the whole Swedish population with diagnostics and expert advice on IEM and has a broad arsenal of biochemical investigations designed to detect defects in intermediary metabolism.

DETAILED DESCRIPTION:
Approximately one in two thousand infants is born with a metabolic disorder that often leads to brain damage. By means of high-tech genetic mapping using whole genome sequencing (WGS), we have discovered the molecular foundations for several of these diseases.

For investigation of mitochondrial diseases, mitochondria are isolated from muscle biopsies for analysis of ATP production using a range of substrate combinations, determination of activities of respiratory chain complexes, and analysis of nuclear and mitochondrial DNA.

The center also performs the national neonatal screening program, currently comprising 26 treatable diseases. Dried blood spot samples (DBS) are stored in the phenylketonuria (PKU) biobank, currently (2024 january) holding around 4.9 million of Sweden's 10.6 million inhabitants.

Many metabolic disorders, however, lack effective counter-measures.

ELIGIBILITY:
Inclusion Criteria:

* Medical inferral, suspicion metabolic disease incl epilepsy and their relatives

Exclusion Criteria:

* Disease other than metabolic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inborn errors of metabolism, a group of around one thousand different monogenic diseases with a wide spectrum of presentation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-04-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetic variant identification using NGS for diagnosis | Through study completion, an average of 1 year.
  Variant identification in patients investigated at our clinic, Centre for inherited metabolic diseases, is an ongoing clinical activity. In many cases, if no variant is identified with NGS (Next Genenation Sequencing) using WGS, additional methods are used such as transcriptomics, proteomics and different cellmodels. More than 400 patients are investigated yearly with NGS/WGS in our clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wedell, Principal Investigator — Karolinska University Hospital, Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No